CLINICAL TRIAL: NCT03044626
Title: Fostering Efficacy of Anti - PD-1 - Treatment: Nivolumab Plus Radiotherapy in Advanced NSCLC
Acronym: FORCE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIO-YMO/TRK-0415; 2015-005741-31 (EudraCT Number); CA209-430 (Other: Bristol-Myers Squibb GmbH & Co. KGaA)
Record Dates: First submitted 2017-01-05; First posted 2017-02-07 (Estimated); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Carcinoma，Non-Small-Cell Lung; Metastatic Lung Cancer; Nonsmall Cell Lung Cancer; Lung Adenocarcinoma Metastatic; Large Cell Lung Carcinoma Metastatic
Keywords: Nivolumab; Radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Radiotherapy; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group A (Experimental): Patients with metastatic non-squamous NSCLC with the necessity of radiotherapy of a metastatic site (e.g. bone) in 2nd-line or 3rd-line treatment:
  Nivolumab 240 mg fixed dose (q2w). First dose followed by radiotherapy. Radiotherapy has to start at the latest 72 hours after nivolumab administration.
  Radiotherapy: A metastatic site will be treated with a radiation dose of 4 Gy for a total of 5 courses during a two week time interval (total dose 20 Gy)
  Interventions: Drug: Radiotherapy; Drug: Nivolumab
- study group B (Other): Patients with metastatic non-squamous NSCLC without the necessity of radiotherapy in 2nd-line or 3rd-line treatment:
  Nivolumab 240 mg fixed dose (q2w).
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Radiotherapy — Nivolumab 240 mg fixed dose (q2w). First dose followed by radiotherapy. Radiotherapy has to start at the latest 72 hours after nivolumab administration.
  Radiotherapy: A metastatic site will be treated with a radiation dose of 4 Gy for a total of 5 courses during a two week time interval (total dose 20 Gy)
  Arms: study group A
Drug: Nivolumab — Nivolumab 240 mg fixed dose (q2w)

SUMMARY:
AIO-YMO/TRK-0415 (FORCE) is a Phase 2, open-label of nivolumab, patients with metastatic non-squamous NSCLC with the necessity of radiotherapy of a metastatic site (e.g. bone) in 2nd-line or 3rd-line treatment for study group A and patients with metastatic non-squamous NSCLC without the necessity of radiotherapy in 2nd-line or 3rd-line treatment for study Group B.

DETAILED DESCRIPTION:
The primary objective is to investigate efficacy of a nivolumab-radiotherapy combination treatment in metastatic non-squamous NSCLC patients.

ELIGIBILITY:
Inclusion criteria

1. Written informed consent and any locally-required authorization (EU Data Privacy Directive in the EU) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations.

2. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

3. Age ≥ 18 years at time of study entry. 4. ECOG performance status 0-1. 5. Patients with measurable disease (at least one uni-dimensionally measurable target lesion by CT-scan or MRI) according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) are eligible. For patients in group A, non-measurable and measurable lesions may be chosen for irradiation. However, in order to allow for evaluation of abscopal effects, patients in group A must have at least one measurable lesion beside the lesion planned to be irradiated. Lesions planned to be irradiated may not be defined as a measurable target lesion. Radiographic tumor assessment must be performed within 28 days before initiation of study treatment.

6. Target Lesions may be located in a previously irradiated field if there is documented (radiographic) disease progression in that site.

7. Patients with metastatic non-squamous non-small cell lung cancer in 2nd-line and 3rd-line treatment and

1. no necessity of radiotherapy or
2. the necessity of radiotherapy of a metastatic bone lesion or soft tissue lesion.

   * Patients with intrathoracic metastases or intrathoracic progressive disease will be included if radiotherapy of the lung parenchyma is NOT required
   * Subjects with symptomatic brain metastases are eligible if metastases have been treated and treatment has been completed at least 12 weeks before inclusion in this study for group B and 2 weeks for group A. Moreover, there must be no magnetic resonance imaging (MRI) evidence of progression within 28 days prior to the first dose of nivolumab administration. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration. Patients with stable/asymptomatic brain metastases that do not require local therapy with irradiation (whole brain irradiation or stereotactic brain irradiation) can be included. In ambiguous cases, consultation with the LKP or his/her delegate is advised.

     8. Patients who will receive study therapy after acceptable prior therapy as specified below are eligible: i. Patients who will receive study therapy as 2nd-line or 3rd-line of treatment:
     1. Patients must have experienced disease recurrence or progression during or after one prior platinum doublet-based chemotherapy regimen for advanced or metastatic disease.

        First line therapy is defined as therapy used to treat advanced disease. Each subsequent line of therapy is preceded by disease progression. A switch of an agent within a regimen in order to manage toxicity does not define the start of a new line of therapy. Subjects must have received at least 2 cycles of platinum doublet based chemotherapy before discontinuation for toxicity.

        Experimental therapies when given as separate regimen are considered as separate line of therapy.

        Maintenance therapy following platinum doublet-based chemotherapy is not considered as a separate regimen of therapy and could comprise continuation of one or more of the agents used in the first-line therapy regimen or switch to another non cross-resistant agent. The initiation of maintenance therapy requires the lack of progressive disease with front-line therapy.

        Treatment given for locally advanced disease is not considered as a line of therapy for advanced disease. Subjects with recurrent disease > 6 months after platinum-containing adjuvant, neoadjuvant or definitive chemoradiation therapy given for locally advanced disease, who also subsequently progressed during or after a platinum doublet-based regimen given to treat the recurrence, are eligible.
     2. Patients who received platinum-containing adjuvant, neoadjuvant or definitive chemoradiation therapy given for locally advanced disease, and developed recurrent (local or metastatic) disease within 6 months of completing therapy are eligible.

        Adjuvant or neoadjuvant platinum-doublet chemotherapy (after surgery and/or radiation therapy) followed by recurrent or metastatic disease within 6 months of completing therapy is considered as first line therapy for advanced disease.

     9. A formalin fixed, paraffin-embedded (FFPE) tumor tissue block (archival or recent) or a minimum of 15 unstained slides of tumor sample (2-3 µm sections, slices must be recent and collected on slides provided by the sponsor) must be available for biomarker (PD-L1) evaluation. Biopsy should be excisional, incisional or core needle. Fine needle aspiration is insufficient.

     10. Prior therapies and surgeries are allowed if completed 2 weeks for minor surgery (group A and B) or 12 weeks for any previous radiotherapy for group B, respectively prior to start of treatment and patient recovered from toxic effects. For group A, any prior radiotherapy not involving the lungs must be completed 2 weeks prior to start of treatment. A prior radiotherapy involving the lungs must be completed 12 weeks prior to start of treatment.

     11. Subjects must have recovered from the effects of major surgery or significant traumatic injury at least 14 days before the first dose of study treatment.

     12. Adequate blood count, liver-enzymes, and renal function (obtained no later than 14 days prior to start of treatment): WBC ≥ 2000/μL Neutrophils ≥ 1500/μL Platelets ≥ 100 x103/μL Hemoglobin ≥ 9.0 g/dL

   Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min (if using the Cockcroft-Gault formula below):

   Female CrCl = ((140 - age in years) x weight in kg x 0.85) / (72 x serum creatinine in mg/dL)

   Male CrCl = ((140 - age in years) x weight in kg x 1.00) / (72 x serum creatinine in mg/dL)

   AST/ALT ≤ 3 x ULN Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)

   13. Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of nivolumab.

   14. Women of childbearing potential must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of nivolumab.

   15. Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product. Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile as well as azoospermic men do not require contraception).

   Exclusion criteria
   1. Previous malignancy (other than NSCLC), which either progresses or requires active treatment.

      Subjects with previous malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colon, cervical/dysplasia, endometrial, melanoma, or breast) are excluded unless a complete remission was achieved at least 2 years prior to study entry AND no additional therapy is required or anticipated to be required during the study period.
   2. Brain metastases mandating active treatment in terms of irradiation (whole brain irradiation or stereotactic brain irradiation). As stated in 3.2 point 7 b, subjects with brain metastases are eligible if metastases have been treated and treatment has been completed at least 12 weeks before inclusion in this study for group B and 2 weeks for group A. Moreover, there must be no magnetic resonance imaging (MRI) evidence of progression within 28 days prior to the first dose of nivolumab administration. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration. Patients with stable/asymptomatic brain metastases that do not require local therapy with irradiation (whole brain irradiation or stereotactic brain irradiation) can be included. In ambiguous cases, consultation with the LKP or his/her delegate is advised.
   3. Known activating EGFR mutation or a known ALK translocation.
   4. Prior therapy with anti-tumor vaccines or other immuno-stimulatory antitumor agents.
   5. Patients with interstitial lung disease.
   6. Any previous treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways
   7. All toxicities attributed to prior anti-cancer therapy other than alopecia and fatigue must have resolved to grade 1 (NCI CTCAE version 4) or baseline before administration of study drug.
   8. Patients should be excluded if they have an active, known or suspected autoimmune disease. NOTE: Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
   9. Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. NOTE: Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
   10. Patients should be excluded if they are positively tested for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection
   11. Patients should be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
   12. History of severe hypersensitivity reactions to other monoclonal antibodies or any excipient.
   13. Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control (failure rate of less than 1% per year)
   14. Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) ≤14 days prior to the first dose of study treatment.
   15. Any other serious or uncontrolled medical disorder, active infection, physical examining, laboratory finding, altered mental status, or psychiatric condition that, in the opinion of the investigator, would limit a subject's ability to comply with the study requirements, substantially increase risk to the subject, or impact the interpretability of study results.
   16. History of solid organ or tissue transplantation including allogenic hematopoietic stem cell transplantation.
   17. Previous enrollment in the present study.
   18. Involvement in the planning and/or conduct of the study (applies to both BMS staff and/or staff of sponsor and study site)
   19. Patient who might be dependent on the sponsor, site or the investigator.
   20. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities § 40 Abs. 1 S. 3 Nr. 4 AMG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
objective response rate (ORR) according to RECIST 1.1 criteria | through study completion, an average of 18 months

SECONDARY OUTCOMES:
progression free survival (PFS) | approx. 6 months
PFS using assessment according to irRECIST | approx. 6 months
  Immune-related Response Evaluation Criteria In Solid Tumors (irRECIST)
ORR using assessment according to irRECIST | approx. 6 months
  Immune-related Response Evaluation Criteria In Solid Tumors (irRECIST)
Overall Survival (OS) | approx. 57 months
Adverse Events | approx. 36 months
  Adverse Events: Type, incidence, and severity according to NCI CTCAE version 4.03
Assesment of Quality of life | approx. 57 months
  as determined with FACT-L (Functional Assessment of Cancer Therapy - Lung)

OTHER OUTCOMES:
Radiation oncology endpoint: absolute size of gross tumor (GTV) | approx. 57 months
Radiation oncology endpoint: clinical target (CTV) | approx. 57 months
Radiation oncology endpoint: planning target volume (PTV) | approx. 57 months
Radiation oncology endpoint: DVH parameters such as D2%, D50%, and D98% within the PTV | approx. 57 months

CONTACTS AND LOCATIONS:
Overall Officials: Farastuk Bozorgmehr, Dr., Principal Investigator — Department of Thoracic Oncology, Thoraxklinik at Heidelberg University Hospital
Locations (16):
- Germany (16):
  - Evangelische Lungenklinik Berlin, Berlin
  - DRK Kliniken Berlin Mitte, Berlin
  - Klinikum Chemnitz, Chemnitz
  - Kliniken der Stadt Köln Krankenhaus Merheim, Cologne
  - Universitätsklinikum Carl-Gustav-Carus, Dresden
  - Klinikum Esslingen GmbH, Esslingen am Neckar
  - Krankenhaus Nordwest, Frankfurt am Main
  - LungenClinic Grosshansdorf, Großhansdorf
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum des Saarlandes, Homburg/Saar
  - Klinikverbund Kempten-Oberallgäu, Immenstadt im Allgäu
  - Klinik Löwenstein, Löwenstein
  - Universitätsklinikum Mannheim, Mannheim
  - Asklepios Fachkliniken München-Gauting, München-Gauting
  - Klinikum Nürnberg, Nuremberg
  - Universitätsklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bozorgmehr F, Chung I, Fischer JR, Bischof M, Atmaca A, Wetzel S, Faehling M, Bottke D, Wermke M, Troost EGC, Kropf-Sanchen C, Wiegel T, Schmidt B, Stupavsky A, Engel-Riedel W, Hammer-Hellmig M, Reinmuth N, Manapov F, Grohe C, Krempien R, Schumann C, Sterzing F, Reck M, Wurschmidt F, Fleckenstein J, Petroff A, Henschke S, Behnisch R, Cvetkovic J, Bruckner L, Schwab C, Stenzinger A, Gotze T, Kopp C, Schroder H, Debus J, Christopoulos P, Thomas M, Rieken S. Reconsidering palliative radiotherapy in addition to PD-1 blockade for non-small cell lung cancer: results from the FORCE phase II trial (AIO/YMO-TRK-0415). Clin Exp Metastasis. 2025 Jul 24;42(5):42. doi: 10.1007/s10585-025-10358-x. PMID 40702361
- [Derived] Bozorgmehr F, Hommertgen A, Krisam J, Lasitschka F, Kuon J, Maenz M, Huber PE, Konig L, Kieser M, Debus J, Thomas M, Rieken S. Fostering efficacy of anti-PD-1-treatment: Nivolumab plus radiotherapy in advanced non-small cell lung cancer - study protocol of the FORCE trial. BMC Cancer. 2019 Nov 8;19(1):1074. doi: 10.1186/s12885-019-6205-0. PMID 31703637
- See also: AIO - Working Group for Medical Oncology from the German Cancer Society — http://www.aio-portal.de
- See also: AIO-Studien-gGmbH — http://www.aio-studien-ggmbh.de